CLINICAL TRIAL: NCT01238523
Title: Early Weight-Bearing in the Closed Treatment of Tibial Shaft Fractures in Children
Brief Title: Study of Tibial Shaft Fractures in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles Orthopaedic Hospital (Other)
Responsible Party: Principal Investigator, Mauricio Silva, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OH-001
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2010-05

CONDITIONS: Tibial Shaft Fractures in Children
Keywords: tibia; shaft; fracture; children
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long leg cast in full extension (Experimental): Long leg cast in full extension with instructions to begin immediate weight bearing as tolerated on the injured extremity
  Interventions: Procedure: Long leg cast in full extension
- Long leg cast with 45 degrees of flexion (Experimental): Long leg cast with 45 degrees of flexion at the knee with instructions not to bear weight on the injured extremity
  Interventions: Procedure: Long leg cast with 45 degrees of flexion

INTERVENTIONS:
Procedure: Long leg cast in full extension — Long leg cast in full extension with instructions to begin immediate weight bearing as tolerated on the injured extremity
  Arms: Long leg cast in full extension
Procedure: Long leg cast with 45 degrees of flexion — Long leg cast with 45 degrees of flexion at the knee with instructions not to bear weight on the injured extremity
  Arms: Long leg cast with 45 degrees of flexion

SUMMARY:
Tibial shaft fracture is one of the most common fractures in children and adolescents. It encompasses approximately 15 % of all long-bone fractures and is third behind only fractures of the femur and both bones of the forearm. (2). Although most authorities agree that closed tibial shaft fractures are best treated by immobilization in a long-leg cast, there is no clear consensus as to when to allow weight bearing on the injured extremity. While most recent articles have recommended long-leg casts with the knee bent in flexion of 30-60 degrees to preclude weight-bearing(1,2,3,4), other authors have recommended much less flexion, 0-5 degrees, to encourage early weight bearing.(5).

The purpose of this randomized controlled prospective study is to determine if the position of immobilization of the knee influences the rate of healing, delayed union, and nonunion As well, we will assess if the type of immobilization affects the function of the patient during the period of treatment using the Activities Scale for Kids - Performance (ASK-P) child self-report musculoskeletal outcome measure . A minimum of 36 patients in each group for a total of 72 patients between 4 and 14 years of age (open physis) with closed fractures of the tibia, with or without fracture of the fibula, will be included in the study

ELIGIBILITY:
Inclusion Criteria:

* Patients between 4 and 14 years of age (open physis)
* Patients seen at the Los Angeles Orthopaedic Medical center within 7 days of the original injury
* All closed tibia and tibia and fibula shaft fractures regardless of fracture pattern

Exclusion Criteria:

* Fractures with greater than 2 cm of initial shortening
* Open fractures
* Patients that have other orthopaedic medical issues such as hemophilia

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The Activities Scale for Kids - Performance (ASK-P) | May 2007 - May 2010
  The Activities Scale for Kids (ASK) is a 30 item child self-report musculoskeletal outcome measure that focuses on the child's physical disability, and is scored with a summary score with no sub-scales. The performance format ASK-P will be used in this study. The scoring system is from 0-100 with 100 being the best possible score.

SECONDARY OUTCOMES:
Time to Healing | May 2007 - May 2010
  Radiographic union will be defined as the presence of callus bridging of 3 out of 4 cortices as seen on anterior posterior and lateral radiographs.

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles Orthopaedic Hospital, Los Angeles, California, United States

REFERENCES:
- [Result] Silva M, Eagan MJ, Wong MA, Dichter DH, Ebramzadeh E, Zionts LE. A comparison of two approaches for the closed treatment of low-energy tibial fractures in children. J Bone Joint Surg Am. 2012 Oct 17;94(20):1853-60. doi: 10.2106/JBJS.J.01728. PMID 23079877